CLINICAL TRIAL: NCT06827977
Title: A Study of Microbiome Transplantation for the Treatment of Constipation and/or Significant Bloating in Patients With Systemic Sclerosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Zsuzsanna Hortobagyi Mcmahan, Associate Professor of Medicine, Co-Director of the UTHealth Scleroderma Center, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-24-0630
Record Dates: First submitted 2025-02-09; First posted 2025-02-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Constipation; Bloating
Keywords: Systemic Sclerosis
MeSH Terms: conditions — Constipation; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PRIM-DJ2727 (Experimental)
  Interventions: Drug: PRIM-DJ2727
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRIM-DJ2727 — For oral administration, each dose will contain the number of capsules needed to deliver the lyophilized intestinal bacteria powder derived after lyophilization of 60 g of filtered stool in 300 mL 0.85% NaCl and 2% mannitol. Participants will take the capsules (5-6 capsules twice weekly) from week 2 through week 10. Capsules will be taken over a period of up to one hour to maximize tolerance and ensure the capsules are not expelled by vomiting.
  For administration via retention enema, which will be done at baseline and week 11, 50 g of filtered, frozen stool in 250 mL of 0.85% sodium chloride (NaCl) will be used.
  Arms: PRIM-DJ2727
Drug: Placebo — Placebo will be administered as capsules from week 2-10 and as enema at baseline and week 11.
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the intestinal flora in subjects with systemic sclerosis-related constipation and/or significant bloating and to determine safety and trends in improvements in the diversity of colonic microbiome and patient symptoms following the administration of either frozen or lyophilized PRIM-DJ2727 microbiota.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the tolerability and safety of frozen and lyophilized microbiome transplant product (PRIM- DJ2727), to characterize the microbiome (α-diversity and β-diversity) and metabolome in patients with Systemic Sclerosis (SSc)-related constipation and/or significant bloating, to examine improvement in constipation and/or significant bloating after microbiome transplant, to examine improved colonic transit after microbiome transplant, to examine subjective global improvement and improvement in SSc disease characteristics, to monitor change in concentration of systemic and fecal inflammatory markers, and to monitor for change in fecal short-chain fatty acids and metabolome.

ELIGIBILITY:
Inclusion Criteria:

* Are seen in the UT Houston Scleroderma Center (UTHSC)
* Meet 2013 American college of rheumatology (ACR)/European league against rheumatism (EULAR) criteria or CREST criteria for SSc
* Meet Rome IV criteria for constipation and/or significant bloating
* Subject willing to sign an informed consent form
* Subject deemed likely to survive for ≥ 1 year after enrollment
* Able to follow study procedure and follow-up
* Sexually active male and female subjects of childbearing potential must agree to use an effective method of birth control during the treatment and follow-up period
* Female subjects of childbearing potential must have a negative pregnancy test in the 72 hours before the procedure
* Subjects who agree to adhere to a stable diet for at least 4 weeks before joining the study and throughout the study
* Subjects must have an attending physician who will provide non-transplant care for the subject

Exclusion Criteria:

* Subjects with constipation and/or significant bloating from causes not attributed to SSc as determined by the treating physician (e.g., inflammatory bowel disease, medication, significant diabetes, or hypothyroidism, etc.)
* Subjects unwilling to stop taking probiotic supplements during the duration of the study
* Subjects that have post-total or hemicolectomy or the presence of a colostomy
* Subjects unable to tolerate microbiome transplant via enema for any reason or swallow capsules
* Subjects requiring systemic antibiotic therapy 4 weeks before the study
* If subjects are on immunosuppression, the immunosuppression dose should be stable for at least 4 weeks before study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms and signs of constipation and/or significant bloating as assessed by total score on the University of California, Los Angeles Gastrointestinal Tract Questionnaire, version 2.0 (UCLA GIT 2.0) | pre-transplant , post-treatment at week 12
  This consists of 34 questions covering domains such as diarrhea, constipation, abdominal pain, nausea, bloating, gastroesophageal reflux, fecal incontinence, and emotional well-being related to GI symptoms. Each item is scored on a Likert scale ranging from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe), with higher scores indicating greater symptom severity. Domain scores are calculated as the sum of responses to items within the domain, and a total score is calculated by summing all domain scores, representing the overall GI symptom burden. Total score will be reported, and the total score ranges from 0-102.
Change in Pelvic Floor Distress as Assessed by the Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20 summary score) | pre-transplant , post-treatment at week 12
  The Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) is composed of 3 subscales: the Urinary Distress Inventory-6 (UDI-6), the Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory-8 (CRADI-8). For each question, the participant must indicate how much bowl, bladder, or pelvic symptoms have been bothering them in the past 3 months on a 4-point scale that ranges from "not at all" (0) to "quite a bit" (4). Total score for each subscale ranges from 0 to 100, with a higher score indicating worse distress. The sum of the 3 subscales are added together to get the PFDI-20 summary score, which ranges from 0 to 300, with a higher score indicating worse distress.
Change in Pelvic Floor Distress as Assessed by the Pelvic Floor Distress Inventory Questionnaire-20 (UDI-6 subscale score) | pre-transplant , post-treatment at week 12
  The Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) is composed of 3 subscales: the Urinary Distress Inventory-6 (UDI-6), the Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory-8 (CRADI-8). For each question, the participant must indicate how much bowl, bladder, or pelvic symptoms have been bothering them in the past 3 months on a 4-point scale that ranges from "not at all" (0) to "quite a bit" (4). Total score for each subscale ranges from 0 to 100, with a higher score indicating worse distress. The sum of the 3 subscales are added together to get the PFDI-20 summary score, which ranges from 0 to 300, with a higher score indicating worse distress.
Change in Pelvic Floor Distress as Assessed by the Pelvic Floor Distress Inventory Questionnaire-20 (POPDI-6 subscale score) | pre-transplant , post-treatment at week 12
  The Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) is composed of 3 subscales: the Urinary Distress Inventory-6 (UDI-6), the Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory-8 (CRADI-8). For each question, the participant must indicate how much bowl, bladder, or pelvic symptoms have been bothering them in the past 3 months on a 4-point scale that ranges from "not at all" (0) to "quite a bit" (4). Total score for each subscale ranges from 0 to 100, with a higher score indicating worse distress. The sum of the 3 subscales are added together to get the PFDI-20 summary score, which ranges from 0 to 300, with a higher score indicating worse distress.
Change in Pelvic Floor Distress as Assessed by the Pelvic Floor Distress Inventory Questionnaire-20 (CRADI-8 subscale score) | pre-transplant , post-treatment at week 12
  The Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) is composed of 3 subscales: the Urinary Distress Inventory-6 (UDI-6), the Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory-8 (CRADI-8). For each question, the participant must indicate how much bowl, bladder, or pelvic symptoms have been bothering them in the past 3 months on a 4-point scale that ranges from "not at all" (0) to "quite a bit" (4). Total score for each subscale ranges from 0 to 100, with a higher score indicating worse distress. The sum of the 3 subscales are added together to get the PFDI-20 summary score, which ranges from 0 to 300, with a higher score indicating worse distress.
Change in symptoms and signs of constipation as assessed by score on the Patient Assessment of Constipation Symptoms (PAC-SYM) scale | pre-transplant , post-treatment at week 12
  The PAC-SYM is a 12-item questionnaire that assesses abdominal, rectal, and stool symptoms, with each item scored from 0 (No symptoms) to 4 (Very severe symptoms), for a total score range of 0-48, with a higher score indicating worse constipation severity.
Change in Gastrointestinal Symptom Severity as Assessed by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) | pre-transplant , post-treatment at week 12
  Total score ranges from 0 (none or absent) to 5 (very severe), with a higher score indicating a worse outcome.
Number of participants who show an improvement in constipation and/or significant bloating symptoms as indicated by the stool diary | from baseline to end of study (week 12)
Change in gut transit times (assessed by Sitz markers and X-ray) | pre-transplant , post-treatment at week 12

SECONDARY OUTCOMES:
Change in immunoglobulin A (IgA) antibody sequence | pre-transplant , week 12 post-transplant
Change in alpha diversity of the microbiome | pre-transplant , week 12 post-transplant
  Species richness and evenness within a single sample will be measured.
Change in beta diversity of the microbiome | pre-transplant , week 12 post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Zsuzsanna McMahan, MD, MHS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No